CLINICAL TRIAL: NCT04340180
Title: Evaluating the Performance of AI in Evaluating Breast MRI Performed With Dose Reduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Stefanie A. Woodard, Assistant Program Director, Diagnostic Radiology Residency Program Assistant Professor, Breast Imaging Section, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R19-159; 000527412 (Other Grant/Funding Number: Bracco)
Record Dates: First submitted 2020-03-31; First posted 2020-04-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Benign Tumor; Breast Malignant Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care; Artificial Intelligence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with enhancing breast lesions (Experimental)
  Interventions: Drug: Standard of Care (SOC) gadolinium Breast MRI; Drug: reduced 1/4 dose gadolinium Breast MRI with Artificial Intelligence (AI) to aid in evaluation.

INTERVENTIONS:
Drug: Standard of Care (SOC) gadolinium Breast MRI — Standard of Care (SOC) gadolinium Breast MRI
Drug: reduced 1/4 dose gadolinium Breast MRI with Artificial Intelligence (AI) to aid in evaluation. — reduced 1/4 dose gadolinium Breast MRI with Artificial Intelligence (AI) to aid in evaluation.

SUMMARY:
The purpose of this study is to evaluate the ability of AI to correctly aid in characterization of benign and malignant lesions even when a low dose of gadolinium is administered. This study is relevant for several reasons, most notably being the reduction of MRI dose and decreased gadolinium deposition in the brain. In addition, use of AI may provide increased sensitivity and specificity for the radiologist evaluating a breast MRI exam. Half of the population will have benign pathologies and the other half will have malignant pathologies.

DETAILED DESCRIPTION:
The study involves each patient presenting for an initial MRI with a regular dose of gadolinium and then presenting at least 48 hours after (no less than 14 days later) for a ¼ dose (see below regarding dosing) gadolinium MRI exam. Both exams will be performed on a 1.5 Tesla magnet. Both exams will include a full protocol. The full dose contrast exam will be read as standard protocol. All images will be anonymized. Images from the reduced dose study will be collected and an AI algorithm applied. All three anonymized data sets (regular dose, low dose, and AI algorithm applied to low dose) will be provided to the readers.

Readers will be three attending radiologists specializing in breast imaging. Exams will be scored on quality, background parenchymal enhancement (BPE), and lesion conspicuity. Enhancing lesions will be identified and characterized by the radiologists in a document provided.

ELIGIBILITY:
Inclusion Criteria for Breast Cancer Patients:

* Female patient between ≥ 18 years old and ≤ 99 years old
* Patients with newly diagnosed primary breast cancer
* Patient able and willing to participate in the trial

Inclusion criteria for Non-malignant indications:

* Female patients between ≥ 18 years old and ≤ 99 years old
* Be referred for MRI for non-malignant indications (screening or BIRADS 3)
* Patients have had prior exam with known enhancing mass, nonmass enhancement, or focus/foci.

Exclusion Criteria:

* Non-female patients
* Patients < 18 years old
* Women who are lactating or pregnant
* Patients with recurrent breast cancer
* Patients who have already received neoadjuvant chemotherapy
* Unable to lie still on the imaging table for one (1) hour
* Patients that are unable to undergo MRI evaluation for reasons specific to MRI

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Compare lesion conspicuity on a scale of 1-4 from low-dose and SOC-dose imaging. | From 1st SOC breast MRI to 2nd low-dose Breast MRI (48 hours to 14 days later).
Compare lesion size in millimeters from low-dose to SOC-dose imaging. | From 1st SOC breast MRI to 2nd low-dose Breast MRI (48 hours to 14 days later).
Compare lesion margins on a scale from 1-4 from low-dose and SOC-dose imaging. | From 1st SOC breast MRI to 2nd low-dose Breast MRI (48 hours to 14 days later).
Compare lesion internal enhancement pattern on a scale from 1-4 from low-dose and SOC- dose imaging. | From 1st SOC breast MRI to 2nd low-dose Breast MRI (48 hours to 14 days later).

SECONDARY OUTCOMES:
Compare the overall background enhancement (scale per standard imaging guidelines. Minimal, mild, moderate, marked). | From 1st SOC breast MRI to 2nd low-dose Breast MRI (48 hours to 14 days later).

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Woodard, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.